CLINICAL TRIAL: NCT00666718
Title: A Prospective Randomized Trial to Compare Basal Bolus Therapies That Use Either Insulin Lispro Protamine Suspension or Insulin Glargine Together With Lispro Insulin in Patients With Type 2 Diabetes
Brief Title: A Comparison Study of Basal Bolus Therapies Together With Lispro Insulin in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12047; F3Z-EW-IOPJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glargine (Active Comparator): Glargine plus Insulin Lispro (2-3 injections)
  Interventions: Drug: Insulin Glargine; Drug: Insulin Lispro
- ILPS (Experimental): Insulin Lispro Protamine Suspension (ILPS) plus Insulin Lispro (2-3 injections)
  Interventions: Drug: Insulin Lispro Protamine Suspension (ILPS); Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Glargine — patient glucose-level dependent, injection, once daily in the evening, 24 weeks
  Arms: Glargine
Drug: Insulin Lispro Protamine Suspension (ILPS) — patient glucose-level dependent, injection, once daily in the evening, 24 weeks
  Other Names: LY275585
  Arms: ILPS
Drug: Insulin Lispro — subcutaneous injections prior to meals, 24 weeks

SUMMARY:
This study is designed to look at if a basal bolus regimen of insulin lispro protamine suspension (ILPS) provides the same glycemic control as a basal bolus regimen of insulin glargine (when one basal bolus regimen is injected once daily together with insulin lispro injected 2-3 times daily).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type 2
* Have been receiving metformin and at least one other oral antihyperglycemic medication (sulfonylurea or thiazolidinedione) with insulin for at least 3 months prior to Visit 1 (Screening)
* Hemoglobin A1C (HbA1c) greater than or equal to 7.5% and less than or equal to 11.0%
* Body Mass Index (BMI) greater than or equal to 25 and less than or equal to 45 kg/m^2
* Capable and willing to follow the protocol
* Give written consent

Exclusion Criteria:

* Are taking any glucose-lowering agents (other than those listed in the inclusion criteria above)
* Have a history of severe hypoglycemia in the past 6 months
* Are pregnant or may become pregnant
* Women who are breastfeeding
* Have significant cardiac disease
* Have significant renal or liver disease
* Undergoing therapy for a malignancy
* Contraindications to the study medications
* Have an irregular sleep/wake cycle
* Have a serious disease or any condition considered by the investigator to be exclusionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willebroek
- Czechia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hranice I-Mesto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olomouc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pilsen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Mergentheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Damme
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pirna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotenburg-Fulda
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ancona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pistoia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ravenna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gorzów Wielkopolski
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mielec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sf Gheorghe
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banská Bystrica
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Modra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nitra
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bornova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, South Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rugby, Warwickshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Bromwich, West Midlands

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Glargine: Glargine plus Insulin Lispro (2-3 injections) plus metformin
- ILPS: Insulin Lispro Protamine Suspension plus Insulin Lispro (2-3 injections) plus metformin
Period: Overall Study
Arm/Group | Glargine | ILPS
Started | 187 | 187
Completed | 175 | 169
Not Completed | 12 | 18
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Entry Criteria Not Met | 2 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine | ILPS | Total
Number analyzed (Participants) | 187 | 187 | 374
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.07) | 59.3 (8.36) | 59.8 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 111 | 212
  Male | 86 | 76 | 162
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 186 | 186 | 372
  African | 0 | 1 | 1
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 5 | 2 | 7
  Czech Republic | 42 | 35 | 77
  Germany | 22 | 20 | 42
  United Kingdom | 10 | 2 | 12
  Greece | 12 | 15 | 27
  Italy | 19 | 26 | 45
  Poland | 32 | 43 | 75
  Romania | 15 | 25 | 40
  Slovakia | 22 | 12 | 34
  Turkey | 8 | 7 | 15
Number of Insulin Injections/Inhalations Per Day [Number; unit: Participants] — The number of insulin injections/inhalations is calculated as the sum of injections per day from the most recently applied insulins before randomization.
  Participants
    1 Insulin Injection/Inhalation per day | 104 | 106 | 210
    2 Insulin Injections/Inhalations per day | 31 | 34 | 65
    3 Insulin Injections/Inhalations per day | 30 | 32 | 62
    4 Insulin Injections/Inhalations per day | 16 | 14 | 30
    >=5 Insulin Injections/Inhalations per day | 6 | 0 | 6
    Missing Data | 0 | 1 | 1
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 93.53 (17.168) | 90.60 (17.075) | 92.06 (17.161)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 33.27 (5.040) | 33.00 (5.004) | 33.13 (5.017)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin] | 8.83 (0.896) | 8.82 (0.895) | 8.82 (0.894)
Duration of Diabetes [Mean (Standard Deviation); unit: Years] | 12.7 (7.04) | 11.8 (6.66) | 12.3 (6.86)
Previous Insulin Treatment [Mean (Standard Deviation); unit: Units (IU)] — The dose is calculated as the total dose from the most recently applied previous insulins before randomization.
  Units (IU) | 36.9 (25.65) | 37.6 (25.75) | 37.3 (25.67)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) to Week 24
Description: Least Squares Mean (LSMean) values reported in the table were controlled for treatment, country, and baseline HbA1c value.
Time Frame: Baseline, Week 24
Population: Per-Protocol Population: All enrolled participants who were randomized and met the following criteria: no violations of Inclusion/Exclusion Criteria have not discontinued study prior to Week 24, compliant as assessed by investigator, and have not been on systemic glucocorticoid therapy for more than 14 consecutive days.
Measure: Least Squares Mean (Standard Error); unit: Percent of Glycosylated Hemoglobin
Groups:
- Glargine: Glargine plus Insulin Lispro (2-3 injections) plus metformin. Participant glucose-level dependent, injection, once daily in the evening, 24 weeks
- ILPS: Insulin Lispro Protamine Suspension plus Insulin Lispro (2-3 injections) plus metformin. Patient glucose-level dependent, injection, once daily in the evening, 24 weeks
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 163 | 148
Percent of Glycosylated Hemoglobin | -1.28 (0.08) | -1.18 (0.09)
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Non-Inferiority or Equivalence — Assuming a drop-out rate after randomization of approximately 15%, the remaining 160 patients in each treatment group should allow confirmation of noninferiority with no true treatment difference and a noninferiority limit of 0.4% using the upper limit of a 2-sided 95% confidence interval ("insulin lispro protamine suspension + insulin lispro" minus "insulin glargine+insulin lispro") at a significance level of 0.025 with 90% power; ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.11 to 0.31]

2. Secondary Outcome: Change From Baseline in HbA1c at Week 12 and Week 24
Description: LSMean values presented were controlled for treatment, country, baseline HbA1C value and week.
Time Frame: Baseline, Week 12, Week 24
Population: Full Analysis Set: All participants who enrolled in this study, were randomized to 1 of the study treatments, and had at least 1 post baseline measurement for the dependent variable, according to intent-to-treat (ITT) principles.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of Glycosylated Hemoglobin
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 180 | 179
Percent of Glycosylated Hemoglobin
  Week 12 Change (n=172, n=168) | -0.99 [-1.14 to -0.84] | -0.90 [-1.10 to -0.69]
  Week 24 Change (n=170, n=166) | -1.29 [-1.45 to -1.13] | -1.07 [-1.28 to -0.86]
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.4580, Mixed Models Analysis — p-value is for Week 12 Change; Change from baseline=Treatment+country+baseline HbA1c+week+treatment*country+treatment*week+baseline HbA1c*treatment (unstructured covariance used)
Statistical Analysis 2: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.1070, Mixed Models Analysis — p-value is for Week 24 Change; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With HbA1c Less Than 7.0% and Less Than or Equal to 6.5% at Endpoint
Time Frame: Week 24
Population: Full Analysis Set: All patients who enrolled in this study, were randomized to 1 of the study treatments, and had at least 1 post baseline measurement for the dependent variable, according to intent-to-treat (ITT) principles.
Measure: Number; unit: Percent of Participants
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 180 | 179
Percent of Participants
  HbA1c < 7.0% | 50 | 36
  HbA1c <= 6.5% | 24 | 14
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.1333, Fisher Exact — p-value is for HbA1c <7.0%
Statistical Analysis 2: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.1213, Fisher Exact — p-value is for HbA1c <=6.5%

4. Secondary Outcome: 7-point Self-monitored Blood Glucose Profiles (SMBG) at Endpoint
Description: LSMean values presented were controlled for treatment, country, and baseline HbA1C value. SMBG at morning pre-meal, morning postprandial, midday pre-meal, midday postprandial, evening pre-meal, evening postprandial, 0300 hours. Postprandial glucose is measured 2 hours after the start of the meal.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 180 | 179
millimoles per liter (mmol/L)
  Morning Pre-Meal | 8.26 (0.22) | 8.63 (0.34)
  Morning Postprandial | 8.93 (0.25) | 9.19 (0.40)
  Midday Pre-Meal | 8.19 (0.23) | 7.90 (0.37)
  Midday Postprandial | 9.11 (0.25) | 9.58 (0.40)
  Evening Pre-Meal | 8.80 (0.24) | 8.75 (0.38)
  Evening Postprandial | 9.27 (0.24) | 9.73 (0.37)
  0300 Hours | 8.16 (0.22) | 8.30 (0.35)
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Morning Pre-Meal measurement = Treatment+country+week+treatment*country + treatment*week (unstructured covariance was used); LS Mean Difference = 0.37, 95% CI 2-sided [-0.43 to 1.17]
Statistical Analysis 2: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Morning Postprandial measurement = Treatment +country+week+treatment*country + treatment*week (unstructured covariance was used); LS Mean Difference = 0.26, 95% CI 2-sided [-0.66 to 1.19]
Statistical Analysis 3: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Midday Pre-Meal measurement = Treatment +country + week +treatment*country + treatment*week (unstructured covariance was used); LS Mean Difference = -0.29, 95% CI 2-sided [-1.15 to 0.57]
Statistical Analysis 4: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Midday Postprandial measurement = Treatment+country+week+treatment*country + treatment*week (unstructured covariance was used); LS Mean Difference = 0.47, 95% CI 2-sided [-0.46 to 1.40]
Statistical Analysis 5: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Evening Pre-Meal measurement = Treatment +country+week+treatment*country + treatment*week (unstructured covariance was used); LS Mean Difference = -0.05, 95% CI 2-sided [-0.93 to 0.83]
Statistical Analysis 6: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Evening Postprandial measurement = Treatment+country+week +treatment*country + treatment*week (unstructured covariance was used); LS Mean Difference = 0.46, 95% CI 2-sided [-0.41 to 1.34]
Statistical Analysis 7: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; 0300 Hours measurement = Treatment+country+week+treatment*country+treatment*week (unstructured covariance was used); LS Mean Difference = 0.14, 95% CI 2-sided [-0.67 to 0.96]

5. Secondary Outcome: Glycemic Variability at Endpoint
Description: LSMeans were controlled for treatment and country grouping (Mediterranean, rest of Europe). Glycemic variability was assessed as the standard deviations of 4 fasting SMBG samples, 4 post-breakfast measurements, 4 post-lunch measurements, 4 post-evening meal measurements.
Time Frame: Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 180 | 179
mmol/L
  Fasting | 0.86 (0.10) | 0.95 (0.10)
  Post-breakfast | 1.56 (0.17) | 1.64 (0.18)
  Post-lunch | 1.61 (0.15) | 1.51 (0.16)
  Post-dinner | 1.43 (0.17) | 1.40 (0.17)
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.5568, ANCOVA — p-value is for Fasting; Glycemic variability = Treatment+country grouping (Mediterranean, rest of Europe)+treatment*country (Mediterranean, rest of Europe)
Statistical Analysis 2: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.7523, ANCOVA — p-value is for Post-breakfast; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.6448, ANCOVA — p-value is for Post-lunch; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.9122, ANCOVA — p-value is for Post-dinner; Glycemic variability = Treatment+country grouping (Mediterranean, rest of Europe)+ treatment*country (Mediterranean, rest of Europe)

6. Secondary Outcome: Rate Of All Self-reported Hypoglycemic Episodes
Description: Rate of self-reported hypoglycemic episodes, all, non-nocturnal,and nocturnal, severe, documented ≤3.9 mmol/L and ≤3.0 mmol/L. Rate=episodes/30 days/patient/. Episode=any time a patient has a symptom associated with hypoglycemia or blood glucose level of ≤70 mg/dL,even if not associated with symptoms.Overall=any time post-randomization in the study period. Nocturnal=Episode between bedtime and waking. Non-Nocturnal=Episode between waking and bedtime.Severe:episode in which patient requires assistance,and has glucose <50 mg/dL or prompt recovery after oral carbohydrate, glucagon, or IV glucose.
Time Frame: Baseline through Week 24
Population: Safety population - all participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: episode/30 days/participant
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 187 | 187
episode/30 days/participant
  All reported episodes rate | 1.38 (0.21) | 0.84 (0.26)
  Nocturnal reported episodes rate | 0.19 (0.05) | 0.15 (0.06)
  Non-Nocturnal reported episodes rate | 1.16 (0.20) | 0.71 (0.24)
  Severe reported episodes rate | 0 (0.013) | 0 (0.029)
  Documented <=3.9 millimoles per liter(mmol/L) rate | 0.89 (0.15) | 0.49 (0.18)
  Documented <=3.0 mmol/L rate | 0.13 (0.04) | 0.12 (0.05)
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Hypoglycemia rate per 30 days = Treatment+Country+Week+Treatment*Country+Treatment*Week (unstructured covariance structure was used); LS Mean Difference = -0.53, 95% CI 2-sided [-1.19 to 0.12]
Statistical Analysis 2: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-0.20 to 0.11]
Statistical Analysis 3: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.45, 95% CI 2-sided [-1.06 to 0.16]
Statistical Analysis 4: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.86 to 0.06]
Statistical Analysis 5: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Hypoglycemia rate per 30 days=Treatment+Country+Week+Treatment*Country+Treatment*Week (unstructured covariance structure was used); LS Mean Difference = -0.01, 95% CI 2-sided [-0.14 to 0.12]

7. Secondary Outcome: Percentage of Participants With Self-Reported Hypoglycemic Episodes
Description: Episode=any time a patient feels that he/she is experiencing a sign or symptom associated with hypoglycemia or has a blood glucose level of ≤70 mg/dL, even if not associated with signs,symptoms, or treatment. Overall=any time post-randomization visits in the study period. Nocturnal=Episode that occurs between bedtime and waking. Non-Nocturnal=Episode occurring between waking and bedtime. Severe=episode with symptoms of neuroglycopenia in which patient requires assistance,and has blood glucose value <50 mg/dL or prompt recovery after oral carbohydrate, glucagon, or intravenous glucose.
Time Frame: Baseline through Week 24
Population: Safety population - all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 187 | 187
percentage of participants
  >=1 hypoglycemic episode | 63.6 | 56.1
  >=1 nocturnal hypoglycemic episode | 19.3 | 25.7
  >=1 non-nocturnal hypoglycemic episode | 61.0 | 54.0
  >=1 severe hypoglycemic episode | 0.5 | 1.6
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.1701, Fisher Exact — p-value is for >=1 hypoglycemic episode
Statistical Analysis 2: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.1727, Fisher Exact — p-value is for >=1 nocturnal hypoglycemic episode
Statistical Analysis 3: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.2094, Fisher Exact — p-value is for >=1 non-nocturnal hypoglycemic episode
Statistical Analysis 4: Comparison: Glargine vs ILPS; Test type: Superiority or Other; p = 0.6230, Fisher Exact — p-value is for >=1 severe hypoglycemic episode

8. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: A listing of adverse events is located in the Reported Adverse Event module.
Time Frame: Baseline through Week 24
Population: Safety population - all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 187 | 187
participants
  AEs | 81 | 65
  Serious adverse events (SAE) | 9 | 14

9. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: LSMean values presented were controlled for treatment, country, and baseline HbA1C value.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 187 | 187
Kilograms (kg) | 1.19 (0.27) | 1.03 (0.30)
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; ANCOVA; weight change from baseline = Treatment + country + baseline Hb1Ac + baseline weight + treatment*HbA1c baseline value; LS Mean Difference = -0.16, 95% CI 2-sided [-0.86 to 0.55]

10. Secondary Outcome: Total Daily Insulin Dose at Endpoint
Description: LSMean values presented were controlled for treatment, country, and baseline HbA1C value.
Time Frame: Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 180 | 179
Units | 78.05 (3.15) | 80.23 (4.31)
Statistical Analysis 1: Comparison: Glargine vs ILPS; Test type: Superiority or Other; Mixed Models Analysis; Total daily insulin dose=Treatment+country+week+treatment*country+ treatment*week (unstructured covariance was used); LS Mean Difference = 2.18, 95% CI 2-sided [-8.33 to 12.68]

11. Secondary Outcome: Number of Injections of Insulin at Week 24
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Glargine | ILPS
Number analyzed (Participants) | 141 | 113
Participants
  2 to <3 per day | 8 | 10
  3 to <4 per day | 129 | 102
  ≥4 per day | 4 | 1

ADVERSE EVENTS:
Groups:
- Glargine/Lispro: Glargine plus Insulin Lispro (2-3 injections) plus metformin
- Lispro/Metformin: Insulin Lispro Protamine Suspension plus Insulin Lispro (2-3 injections) plus metformin
Arm/Group | Glargine/Lispro | Lispro/Metformin
Serious Adverse Events (participants affected / at risk) | 9/187 | 14/187
Other Adverse Events (participants affected / at risk) | 81/187 | 65/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine/Lispro (N=187) | Lispro/Metformin (N=187)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — This event resulted in death.
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Oedema mucosal (General disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Physiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine/Lispro (N=187) | Lispro/Metformin (N=187)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 4 (6)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 5 (5) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (17) | 10 (12)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pulpitis dental (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 3 (4) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 5 (7) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 11 (20) | 9 (39)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (7) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Cataract operation (Surgical and medical procedures) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days